CLINICAL TRIAL: NCT02146170
Title: Tissue Procurement and Natural History Study of Patients With Non-Small Cell Lung Cancer, Small Cell Lung Cancer, Extrapulmonary Small Cell Cancer, Pulmonary Neuroendocrine Tumors, and Thymic Epithelial Tumors
Brief Title: Tissue Procurement and Natural History Study of People With Non-Small Cell Lung Cancer, Small Cell Lung Cancer, Extrapulmonary Small Cell Cancer, Pulmonary Neuroendocrine Tumors, and Thymic Epithelial Tumors
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140105; 14-C-0105
Record Dates: First submitted 2014-05-08; First posted 2014-05-23 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-09-17

CONDITIONS: Non-Small Cell Lung Cancer; Small Cell Lung Cancer; Extrapulmonary Small Cell Cancer; Pulmonary Neuroendocrine Tumors; Thymic Epithelial Tumors
Keywords: Sample Acquisition; Genetic and Epigenetic Alterations; Mig6 Expression; Proteomic Analysis; Genomic Analysis; Natural History
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group: Patients with histologically or cytologically confirmed NSCLC, SCLC, ESCC, PNET, and TET

SUMMARY:
Background:

- Lung cancer is the leading cause of cancer-related death worldwide. It causes more than one million deaths every year. Researchers want to gather tissue samples from people with lung and thymic cancers to understand the disease better. This may lead to new ways to diagnose and treat it.

Objective:

- To collect tissue samples for use in the study of lung cancers.

Eligibility:

- Adults over age 18 with non-small cell lung cancer, small cell lung cancer, extra pulmonary small cell cancer, pulmonary neuroendocrine tumors, and thymic epithelial tumors.

Design:

* Participants will be screened with a medical history, physical exam, and blood tests. They will be asked about how they perform their daily tasks.
* Participants may be asked to give urine and blood samples. They may give a saliva sample if they cannot give blood. They will also give a sample of their tumor from a biopsy they had. They may also be given the option to undergo a biopsy.
* Participants may have MRI, CT, and/or PET scans of the body. They will lie in a machine that takes pictures of the body.
* After visits to the Clinical Center end, researchers will contact participants by phone every year to check on their health.

DETAILED DESCRIPTION:
Background:

* Lung cancer is the leading cause of cancer-related death worldwide, accounting for more than one million deaths every year.
* Several genetic and epigenetic alterations are involved in initiation and progression of NSCLC. Some of these alterations are seen in normal and pre-neoplastic cells as well, suggesting a sequential development from normal epithelial cells to cancer, through a multistep process, usually coincident with cigarette smoking.
* This natural history protocol is an extension of our Molecular Profiling protocol to enable tissue collection for more in-depth proteomic and genomic analyses to understand tumor biology and treatment response.
* A cohort of patients enrolled in this natural history study is likely to enroll in the IRB approved protocol for end-of-life in-patient hospice and rapid autopsy following death (13-C-0131). Longitudinally collected tumor tissue from these patients, including from several metastatic sites at autopsy will be a unique resource to understand tumor evolution.
* There will be opportunity to embark upon a wide array of studies in the future with the longitudinally collected tissue samples tagged with clinical information from patients.

Objectives:

- To allow sample acquisition for use in the study of non-small cell lung cancer (NSCLC), Small cell lung cancer (SCLC), extrapulmonary small cell cancer (ESCC), pulmonary neuroendocrine tumors (PNET), and thymic epithelial tumors (TETs).

Eligibility:

* Patients with histologically or cytologically confirmed NSCLC, SCLC, ESCC, PNET, and TET.
* Patients consulted in the Clinical Center without a definitive diagnosis, but clinically considered likely to have a thoracic malignancy of the above histologies, pending further tissue acquisition and/or pathology review.
* Age greater than or equal to 18 years.

Design:

* This is a biospecimen collection and natural history protocol in which samples will be collected from patients with NSCLC, SCLC, ESCC, PNET, and TET.
* Eligible patients undergoing screening for or participating in NIH protocols or eligible patients treated elsewhere and referred from other oncologists will be referred for participation in this study.
* Upon providing informed consent, patients will undergo sample acquisition procedures, which may include a tumor biopsy, bone marrow biopsy or the collection of blood, urine or other body fluids.
* An accrual ceiling of 2000 subjects is planned.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Individuals with histologically or cytologically confirmed NSCLC, SCLC, ESCC, PNET, and TET.
* Individuals consulted in the Clinical Center without a definitive diagnosis, but clinically considered likely to have a malignancy of the above histologies, pending further tissue acquisition and/or pathology review.
* Age greater than or equal to18 years. Children are excluded from the study, as the above thoracic malignancies are rare in this population.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Active symptomatic major organ disorder that would increase the risk of biopsy, including but not limited to ischemic heart disease, recent myocardial infarction, active congestive heart failure, pulmonary dysfunction.
* Active concomitant medical or psychological illnesses that may increase the risk to the subject, at the discretion of the Principal Investigator.
* Known HIV-positive individuals not on combination antiretroviral therapy are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically or cytologically confirmed NSCLC, SCLC, ESCC, PNET, and TET
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-05-28 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Allow sample acquisition for use in the study of thoracic malignancies except mesothelioma. | Ongoing
  blood, tumor, body fluids, and normal tissue samples

SECONDARY OUTCOMES:
Follow the natural history of patients with thoracic malignancies. | ongoing
  clinical data, including overall survival
Conduct genomic, proteomic and immunological analyses on blood, tumor, body fluid and normal tissue in support of NIH translational trials to develop new therapeutic agents and novel treatment approaches as well as new prognostic and diagnostic ... | ongoing
  Specific studies include, but not limited to genomic analyses using NGS technologies (exome, transcriptome and/or whole genome sequencing), DNA methylation analyses, DNA copy number analyses, proteomic studies including mass spectrometry, capillary Westerns, reverse phase protein microarrays (RPPA), luminex assays, ELISA and IHC, and metabolomics studies using mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rajan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Weir BA, Woo MS, Getz G, Perner S, Ding L, Beroukhim R, Lin WM, Province MA, Kraja A, Johnson LA, Shah K, Sato M, Thomas RK, Barletta JA, Borecki IB, Broderick S, Chang AC, Chiang DY, Chirieac LR, Cho J, Fujii Y, Gazdar AF, Giordano T, Greulich H, Hanna M, Johnson BE, Kris MG, Lash A, Lin L, Lindeman N, Mardis ER, McPherson JD, Minna JD, Morgan MB, Nadel M, Orringer MB, Osborne JR, Ozenberger B, Ramos AH, Robinson J, Roth JA, Rusch V, Sasaki H, Shepherd F, Sougnez C, Spitz MR, Tsao MS, Twomey D, Verhaak RG, Weinstock GM, Wheeler DA, Winckler W, Yoshizawa A, Yu S, Zakowski MF, Zhang Q, Beer DG, Wistuba II, Watson MA, Garraway LA, Ladanyi M, Travis WD, Pao W, Rubin MA, Gabriel SB, Gibbs RA, Varmus HE, Wilson RK, Lander ES, Meyerson M. Characterizing the cancer genome in lung adenocarcinoma. Nature. 2007 Dec 6;450(7171):893-8. doi: 10.1038/nature06358. Epub 2007 Nov 4. PMID 17982442
- [Background] Imielinski M, Berger AH, Hammerman PS, Hernandez B, Pugh TJ, Hodis E, Cho J, Suh J, Capelletti M, Sivachenko A, Sougnez C, Auclair D, Lawrence MS, Stojanov P, Cibulskis K, Choi K, de Waal L, Sharifnia T, Brooks A, Greulich H, Banerji S, Zander T, Seidel D, Leenders F, Ansen S, Ludwig C, Engel-Riedel W, Stoelben E, Wolf J, Goparju C, Thompson K, Winckler W, Kwiatkowski D, Johnson BE, Janne PA, Miller VA, Pao W, Travis WD, Pass HI, Gabriel SB, Lander ES, Thomas RK, Garraway LA, Getz G, Meyerson M. Mapping the hallmarks of lung adenocarcinoma with massively parallel sequencing. Cell. 2012 Sep 14;150(6):1107-20. doi: 10.1016/j.cell.2012.08.029. PMID 22980975
- [Background] Rikova K, Guo A, Zeng Q, Possemato A, Yu J, Haack H, Nardone J, Lee K, Reeves C, Li Y, Hu Y, Tan Z, Stokes M, Sullivan L, Mitchell J, Wetzel R, Macneill J, Ren JM, Yuan J, Bakalarski CE, Villen J, Kornhauser JM, Smith B, Li D, Zhou X, Gygi SP, Gu TL, Polakiewicz RD, Rush J, Comb MJ. Global survey of phosphotyrosine signaling identifies oncogenic kinases in lung cancer. Cell. 2007 Dec 14;131(6):1190-203. doi: 10.1016/j.cell.2007.11.025. PMID 18083107
- [Derived] Wong-Rolle A, Dong Q, Zhu Y, Divakar P, Hor JL, Kedei N, Wong M, Tillo D, Conner EA, Rajan A, Schrump DS, Jin C, Germain RN, Zhao C. Spatial meta-transcriptomics reveal associations of intratumor bacteria burden with lung cancer cells showing a distinct oncogenic signature. J Immunother Cancer. 2022 Jul;10(7):e004698. doi: 10.1136/jitc-2022-004698. PMID 35793869
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-C-0105.html